CLINICAL TRIAL: NCT04173221
Title: Direct Assessment of Microcirculation In Shock (DAMIS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: DAMIS
Record Dates: First submitted 2019-11-15; First posted 2019-11-21 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Microcirculation; Intensive Care; Shock
Keywords: Microcirculation; Intensive Care; Critical care; shock; risk stratification; SDF-measurement; fluid resuscitation
MeSH Terms: conditions — Shock

STUDY DESIGN:
Intervention Model Description: Sublingual SDF-Measurement at admission and after 24h, with or without communication and interpreting checklist to the treating physician
Who Masked: Investigator
Masking Description: Sublingual SDF-Measurement at admission and after 24h, with or without communication and interpreting checklist to the treating physician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Sublingual SDF-Measurement with communication and interpreting checklist to the treating physician
- Control (Other)
  Interventions: Other: Sublingual SDF-Measurement without communication and interpreting checklist to the treating physician

INTERVENTIONS:
Other: Sublingual SDF-Measurement with communication and interpreting checklist to the treating physician — Sublingual SDF-Measurement at admission and after 24h, with communication and interpreting checklist to the treating physician
  Arms: Intervention
Other: Sublingual SDF-Measurement without communication and interpreting checklist to the treating physician — Sublingual SDF-Measurement at admission and after 24h, without communication and interpreting checklist to the treating physician
  Arms: Control

SUMMARY:
Maintaining organ perfusion is the key to successful intensive care medicine. Shock is the most dangerous microcirculatory disorder and one of the most hazardous and lethal conditions of critically ill patients still showing high mortality rates. However, there are still ongoing controversies, how to assess microcirculation, how to predict outcome in time and how to guide specific therapy. Macrocirculation does not reflect microcirculation. Microcirculation reflects organ perfusion and correlates with the outcome. There is growing evidence that microcirculatory parameters are powerful tools to predict the outcome after cardiac arrest. Several guidelines use it as a target to guide therapy, but these recommendations base only on supporting evidence of low quality. Lactate is a late reflector of reduced organ perfusion and is of limited value for time-critical decision-making and their value as a therapeutic target. Sublingual sidestream dark-field (SDF) - measurement is a non-invasive method that reliably reflects organ perfusion. The last generation of microcirculation assessment tools are easy to use hand-held devices that use an automatic algorithm. In consequence, microcirculation has become a directly detectable physiological compartment. However, systematic investigations about this technology in shock are still lacking. DAMIS determines the value of directly assessed microcirculation on outcome in different types of shock. Therefore, this multicenter study will recruit up to 200 patients in shock. After the first measurement, patients will be randomized either to intervention or to control. The intervention consists in knowing microcirculatory parameters. A checklist will assist the treating physicians of the interventional group in explaining microcirculatory values and offering possible treatment options. Patients in the control group will be measured as well, but results will not be communicated to the treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years
2. Admitted to the ICU in state of shock at the time point of admission to ICU or in the first 3 hours defined as

   * the need to use vasopressors, -dilatators, fluids to maintain mean arterial pressure > 65 mmHg
   * AND lactate > 2 mmol/l

Exclusion Criteria:

1. Younger than 18 years
2. Anatomic reasons that inhibit sublingual measurement
3. Lack of informed consent
4. more than 4 hours after ICU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-08-27 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
mortality | 30 day
  relationship of bedside measurement of microcirculation with the clinical outcome in terms of mortality

SECONDARY OUTCOMES:
mortality | 6 and 12 months
  relationship of bedside measurement of microcirculation with the clinical outcome in terms of mortality
length of stay at ICU and hospital | 90 days
  relationship of bedside measurement of microcirculation with the clinical outcome in terms of length of stay

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf
  - Department of Anaesthesiology and Critical Care, Medical Centre - University of Freiburg, Faculty of Medicine, Freiburg im Breisgau
  - Department of Anesthesiology, Center of Anesthesiology and Intensive Care Medicine, University Medical Center Hamburg-Eppendorf, Hamburg
  - Department of Cardiology, Heart Center Leipzig at University of Leipzig, Leipzig
  - Robert-Bosch-Krankenhaus, Department of Anesthesiology and Intensive Care Medicine, Stuttgart

REFERENCES:
- [Derived] Bruno RR, Hernandez G, Thiele H, Kattan E, Jung C; DAMIS study group. A microcirculation-guided trial: never trying is worse than failing. Intensive Care Med. 2023 Dec;49(12):1555-1556. doi: 10.1007/s00134-023-07245-y. Epub 2023 Oct 9. No abstract available. PMID 37812227
- [Derived] Bruno RR, Hernandez G, Wollborn J, Saugel B, Jung C; of the DAMIS study group. Microcirculation information in clinical decision making: Rome wasn't built in a day. Intensive Care Med. 2023 Oct;49(10):1272-1273. doi: 10.1007/s00134-023-07216-3. Epub 2023 Sep 11. No abstract available. PMID 37695331
- [Derived] Bruno RR, Wollborn J, Fengler K, Flick M, Wunder C, Allgauer S, Thiele H, Schemmelmann M, Hornemann J, Moecke HME, Demirtas F, Palici L, Franz M, Saugel B, Kattan E, De Backer D, Bakker J, Hernandez G, Kelm M, Jung C. Direct assessment of microcirculation in shock: a randomized-controlled multicenter study. Intensive Care Med. 2023 Jun;49(6):645-655. doi: 10.1007/s00134-023-07098-5. Epub 2023 Jun 6. PMID 37278760